CLINICAL TRIAL: NCT01992614
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of PF-06678552 After Fed And Fasted Administration Of Single Escalating Oral Doses In Healthy Subjects
Brief Title: A Single Dose Study Of PF-06678552 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7611001
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Single Ascending Dose; healthy subjects; Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Single ascending doses of PF-06678552 or placebo to investigate the safety, tolerability, PK, and PD.
  Interventions: Drug: PF-06678552 or Placebo
- Cohort 2 (Experimental): Single ascending doses of PF-06678552 or placebo to investigate the safety, tolerability, PK, and PD.
  Interventions: Drug: PF-06678552 or Placebo
- Cohort 3 (Experimental): Single ascending doses of PF-06678552 or placebo to investigate the safety, tolerability, PK, and PD.
  Interventions: Drug: PF-06678552 or Placebo

INTERVENTIONS:
Drug: PF-06678552 or Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution once in each period.
  Arms: Cohort 1
Drug: PF-06678552 or Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution once in each period.
  Arms: Cohort 2
Drug: PF-06678552 or Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution once in each period.
  Arms: Cohort 3

SUMMARY:
PF-06678552 is a new compound proposed for the treatment of hypercholesteremia. The primary purpose of this study is to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of single oral doses of PF-06678552 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential.
* Body Mass Index (BMI) of 18 to 30.5 kg/m2; and a total body weight >50 kg
* Low density lipoprotein cholesterol between 115 mg/dL and 190 mg/dL

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs), clinical laboratory tests, vital signs (including blood pressure and pulse rate) and cardiac conduction intervals as assessed via 12-lead electrocardiogram (ECG). | 0 to 72 hours post dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06678552 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - infinity)] for PF-06678552 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  AUC (0 - infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Maximum Observed Plasma Concentration (Cmax) for for PF-06678552 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06678552 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) for PF-06678552 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Apparent Oral Clearance (CL/F) for PF-06678552 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) for PF-06678552 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06644927 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - infinity)] for PF-06644927 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  AUC (0 - infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Maximum Observed Plasma Concentration (Cmax) for PF-06644927 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06644927 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) for PF-06644927 | 0, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Amount of PF-06644927 excreted in the urine (Ae) | 0-4, 4-12, and 12-24 hours post dose
  Amount of drug excreted in the urine is a measure of the degree that the kidneys filter drug from the blood to the urine.
Percent of PF-06678552 dose excreted in the urine as PF-06644927 (Ae%) | 0-4, 4-12, and 12-24 hours post dose
  The percent of PF-06678552 dose excreted in the urine as PF-06644927 is calculated from the mass of dose excreted in the urine compared to the total dose of PF-06678552 and corrected for the relative weight of PF-06644927 to PF-06678552.
Renal Clearance (CLr) for PF-06644927 | 0-4, 4-12, and 12-24 hours post dose
  Renal clearance is the measure of the rate of drug moving into the urine from blood

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7611001&StudyName=A%20Single%20Dose%20Study%20Of%20PF-06678552%20In%20Healthy%20Subjects